CLINICAL TRIAL: NCT03270865
Title: Usability and Ergonomic Evaluation of Self-Positioning System for Retinal Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Notal U-001 V. 1.0
Record Dates: First submitted 2017-08-15; First posted 2017-09-01 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: AMD Population - Intermediate or Advanced AMD; DR Population- With or Without Diabetic Macular Edema
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usability and Ergonomic Evaluation of Self-Positioning System (Experimental)
  Interventions: Device: PAF (Positioning And Fixation device)

INTERVENTIONS:
Device: PAF (Positioning And Fixation device) — Up to 60 Subjects will be evaluating for positioning accuracy and comfort by comparing different methods utilizing the PAF device. Some methods of positioning will be applied and compare for each usability factor X, Y, Z location, and fixation.
  The patient will be evaluated before pupil dilation. VA and ophthalmic diagnoses will be recorded.
  Pupil position will be recorded using 3 commercial off the shelf cameras when the subject is performing simple ergonomic tasks while looking at a screen presenting images. Each testing session will be limited 20 min long. Subjects will be able to rest within the testing session if required. Total session time per patient will not exceed 30 minutes.

SUMMARY:
The purpose of the study "Usability and Ergonomic Evaluation of Self-Positioning System for Retinal Imaging" is to enable self-operation of a monitoring device in home-simulated environment

DETAILED DESCRIPTION:
One of the main challenges in developing a retinal imager is to design it to be self-operated by elderly patients in their home setting The study's objective is to explore ergonomic solutions that will allow the user to perform imaging on their own. The study will be done in a home-simulated environment using a dedicated ergonomic system (termed "PAF" - Positioning And Fixation system) that stimulates the retinal imager and enables to record the tested subject using standard cameras. The prototype doesn't include the retinal imager and does not include any imaging capabilities aside from standard means of photography Subjects will be evaluating for positioning accuracy and comfort by comparing different methods. Pupil position will be recorded using commercial off the shelf cameras when the subject is performing simple ergonomic tasks while looking at a screen presenting images.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* Able to understand and sign the informed consent form
* Ability to communicate verbally
* AMD (interim and advanced) or diabetic retinopathy (with and without DME)

Exclusion Criteria:

* Visual acuity >=20/200 in the better eye

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
spatial location of the pupil, during an eye examination | 1 year
  documentation of pupil location by a camera

CONTACTS AND LOCATIONS:
Locations (1):
- Sorasky Medical Center, Tel Aviv, Israel